CLINICAL TRIAL: NCT03697616
Title: Ridge Augmentation Using Autologous Concentrated Growth Factors (CGF) Enriched Bone Graft Matrix (Sticky Bone) Versus Guided Bone Regeneration Using Native Collagen Membrane in Horizontally Deficient Maxilla
Brief Title: Horizontal Maxillary Ridge Augmentation With Sticky Bone Versus Collagen Membrane GBR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah AbdAllah Mohamed, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CairoUImp
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Horizontal Deficiecy in Maxillary Arches

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ridge augmentation with sticky bone and GBR (Experimental): Ridge augmentation using Autologous concentrated Growth factors (CGF) enriched bone graft matrix (sticky bone) and guided bone regeneration using native collagen membrane in horizontally deficient maxilla
  Interventions: Device: Ridge augmentation with sticky bone and GBR

INTERVENTIONS:
Device: Ridge augmentation with sticky bone and GBR — * Autogenous particulate bone will be harvested and a mixture of autogenous particulate and anorganic bovine bone mineral will be prepared at a ratio of 1:1
  * Venous blood will be drawn from patients' forearm and centrifuged at 2500 RPM/3 minutes and 4000 RPM/15 minutes to produce autologous fibrin glue and concentrated growth factors membrane, respectively
  * Sticky bone will be prepared by adding autologous fibrin glue to the particulate mixture, placed onto the defect and covered by the prepared concentrated growth factors membrane
  * For guided bone regeneration the particulate mixture will be placed onto the defect and covered by resorbable collagen membrane
  * Periosteal releasing incision will be done to provide flap advancement for tension free closure
  * Closure will be done using horizontal mattress and interrupted 4/0 polypropylene sutures

SUMMARY:
Guided bone regeneration (GBR) using bone graft and barrier membrane is a well-established technique for augmentation of atrophic alveolar ridges. There are many techniques for ridge augmentation involves the use of bone grafting materials, barrier membranes, possibly some tenting/fixation screws the stability of bone graft, space maintenance, angiogenesis, and tension free primary suture are essential for success.

DETAILED DESCRIPTION:
Common techniques introduced for horizontal ridge augmentation are Guided Bone Regeneration (GBR), there are many techniques for ridge augmentation involves the use of bone grafting materials, barrier membranes, possibly some tenting/fixation screws. For successful GBR, stability of bone graft, space maintenance, angiogenesis, and tension free primary suture are essential. Space maintenance with particulate bone graft should be provided during healing period. However particulate bone graft is easily migrated when grafted on the large horizontal bone defect. To reconstruct large bony defect or for the 3-dimensional ridge augmentation, bone tack on the collagen membrane or titanium mesh is required to contain particulate bone graft during healing but these procedures are surgically time consuming and technique sensitive.

Sticky bone is biologically solidified bone graft which is entrapped in fibrin network. Sticky bone graft doesn't scatter because particulate bone powders are strongly interconnected each other by fibrin network.

ELIGIBILITY:
Inclusion Criteria:

* Inadequate facial bone obviating prosthodontically planned implant placement in the maxilla
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement.

Exclusion Criteria:

* Significant bone-related illness or pathology.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia, or bone augmentation to implant site
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone gain | 6 months
  The amount of horizontal bone gain will be measured by cone beam computed tomography